CLINICAL TRIAL: NCT00633373
Title: An Open-label Treatment Use Protocol of Cyclosporine Inhalation Solution (CIS) in Lung Transplant Recipients
Brief Title: Cyclosporine Inhalation Solution (CIS) in Lung Transplant Recipients
Status: No longer available | Type: Expanded Access
Sponsor: APT Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ACS004
Record Dates: First submitted 2008-03-05; First posted 2008-03-12 (Estimated); Last update posted 2012-09-17 (Estimated); Status verified 2012-09

CONDITIONS: Lung Transplant
Keywords: lung; transplant; transplant rejection; Cyclosporine; bronchiolitis obliterans; aerosol
MeSH Terms: conditions — Bronchiolitis Obliterans

INTERVENTIONS:
Drug: Cyclosporine Inhalation Solution — Cyclosporine USP Inhalation Solution (CIS) 300mg/4.8 mL delivered via a disposable nebulizer. A titration phase of 10 days is recommended starting with 100 mg and then increasing over the 10 days to a maximum of 300 mg or the highest tolerated dose.

SUMMARY:
Currently there are no approved therapies for lung transplant recipients in the United States (US). Treatment with CIS following lung transplantation has previously been demonstrated to result in a clinically meaningful improvement in survival and chronic rejection-free survival compared to placebo, but additional data supporting its use is needed prior to Food and Drug Administration (FDA) approval. This treatment use protocol is a mechanism for providing eligible lung transplant recipients early access to CIS in advance of FDA approval.

ELIGIBILITY:
Inclusion Criteria:

* Single-or double-lung transplant recipients who have a high risk for developing chronic rejection
* Single or double-lung transplant recipients who have developed chronic rejection
* Single or double-lung transplant recipients who have serious or life-threatening complications of systemic immunosuppressive therapy

Exclusion Criteria:

* Known hypersensitivity to cyclosporine or propylene glycol (PG)
* Females who are pregnant or are considering becoming pregnant
* Females who are breast feeding a child.

Sex: All
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - University of California at San Francisco, San Francisco, California
  - University of Florida Health Sciences Center, Gainesville, Florida
  - Tampa General Hospital, Tampa, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Children's Hospital Boston, Boston, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor Clinic, Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Background] Burkart GJ, Smaldone GC, Eldon MA, Venkataramanan R, Dauber J, Zeevi A, McCurry K, McKaveney TP, Corcoran TE, Griffith BP, Iacono AT. Lung deposition and pharmacokinetics of cyclosporine after aerosolization in lung transplant patients. Pharm Res. 2003 Feb;20(2):252-6. doi: 10.1023/a:1022275222207. PMID 12636164
- [Background] Iacono AT, Smaldone GC, Keenan RJ, Diot P, Dauber JH, Zeevi A, Burckart GJ, Griffith BP. Dose-related reversal of acute lung rejection by aerosolized cyclosporine. Am J Respir Crit Care Med. 1997 May;155(5):1690-8. doi: 10.1164/ajrccm.155.5.9154878.
- [Background] Keenan RJ, Iacono A, Dauber JH, Zeevi A, Yousem SA, Ohori NP, Burckart GJ, Kawai A, Smaldone GC, Griffith BP. Treatment of refractory acute allograft rejection with aerosolized cyclosporine in lung transplant recipients. J Thorac Cardiovasc Surg. 1997 Feb;113(2):335-40; discussion 340-1. doi: 10.1016/S0022-5223(97)70331-3. PMID 9040628
- [Background] Iacono A, Dauber J, Keenan R, Spichty K, Cai J, Grgurich W, Burckart G, Smaldone G, Pham S, Ohori NP, Yousem S, Williams P, Griffith B, Zeevi A. Interleukin 6 and interferon-gamma gene expression in lung transplant recipients with refractory acute cellular rejection: implications for monitoring and inhibition by treatment with aerosolized cyclosporine. Transplantation. 1997 Jul 27;64(2):263-9. doi: 10.1097/00007890-199707270-00015. PMID 9256185
- [Background] Iacono AT, Johnson BA, Grgurich WF, Youssef JG, Corcoran TE, Seiler DA, Dauber JH, Smaldone GC, Zeevi A, Yousem SA, Fung JJ, Burckart GJ, McCurry KR, Griffith BP. A randomized trial of inhaled cyclosporine in lung-transplant recipients. N Engl J Med. 2006 Jan 12;354(2):141-50. doi: 10.1056/NEJMoa043204. PMID 16407509
- [Background] Iacono AT, Corcoran TE, Griffith BP, Grgurich WF, Smith DA, Zeevi A, Smaldone GC, McCurry KR, Johnson BA, Dauber JH. Aerosol cyclosporin therapy in lung transplant recipients with bronchiolitis obliterans. Eur Respir J. 2004 Mar;23(3):384-90. doi: 10.1183/09031936.04.00058504. PMID 15065826
- [Background] Iacono AT, Keenan RJ, Duncan SR, Smaldone GC, Dauber JH, Paradis IL, Ohori NP, Grgurich WF, Burckart GJ, Zeevi A, Delgado E, O'Riordan TG, Zendarsky MM, Yousem SA, Griffith BP. Aerosolized cyclosporine in lung recipients with refractory chronic rejection. Am J Respir Crit Care Med. 1996 Apr;153(4 Pt 1):1451-5. doi: 10.1164/ajrccm.153.4.8616581.